CLINICAL TRIAL: NCT00027638
Title: Phase II Trial Of Thalidomide In Patients With Low Grade Neuroendocrine Tumors (Carcinoid and Islet Cell Cancers)
Brief Title: Thalidomide in Treating Patients With Metastatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: MSKCC-01027; CDR0000069051 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-2029
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Gastrointestinal Carcinoid Tumor; Islet Cell Tumor; Lung Cancer; Neoplastic Syndrome
Keywords: metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; gastrinoma; insulinoma; recurrent islet cell carcinoma; WDHA syndrome; somatostatinoma; pancreatic polypeptide tumor; glucagonoma; pulmonary carcinoid tumor
MeSH Terms: conditions — Adenoma, Islet Cell; Lung Neoplasms; Neoplasms; Gastrinoma; Insulinoma; Carcinoma, Islet Cell; Vipoma; Somatostatinoma; Glucagonoma | interventions — Thalidomide

INTERVENTIONS:
Drug: thalidomide

SUMMARY:
RATIONALE: Thalidomide may stop the growth of neuroendocrine tumors by stopping blood flow to the tumor.

PURPOSE: Phase II trial to study the effectiveness of thalidomide in treating patients who have metastatic neuroendocrine tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and efficacy of thalidomide in patients with metastatic low-grade neuroendocrine tumors.

OUTLINE: Patients receive oral thalidomide once daily on weeks 1-8. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 14-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed low-grade neuroendocrine tumors

  * Carcinoid tumors
  * Islet cell tumors
* Metastatic disease
* Progression of disease within past 4 weeks by radiological evidence
* At least 1 bidimensionally measurable lesion by CT scan or MRI

  * Bone metastasis not considered measurable if only site of disease
* No active brain metastases

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Karnofsky 70-100%

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* AST no greater than 2.5 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance at least 50 mL/min

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of effective contraception for 4 weeks before, during, and for 4 weeks after study
* No grade 2 or greater neuropathy
* No other clinical circumstances that would preclude study
* No other prior malignancy except:
* Non-melanoma skin cancer
* Other cancer that has been curatively treated, has had no evidence of recurrence within the past 5 years, and is at low risk for recurrence

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior thalidomide
* No concurrent interferon

Chemotherapy:

* No concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* At least 4 weeks since prior major surgery

Other:

* No more than 1 prior systemic therapy regimen
* At least 4 weeks since prior systemic therapy regimen
* No other concurrent therapeutic agent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-03; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard B. Saltz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States